CLINICAL TRIAL: NCT03373305
Title: A Phase 1 Trial of Brentuximab Vedotin Plus Lenalidomide in Patients With Relapsed/ Refractory Cutaneous T-Cell Lymphomas
Brief Title: Brentuximab Vedotin and Lenalidomide in Treating Patients With Relapsed or Refractory T-Cell Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: contract not executed
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17347; NCI-2017-02163 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-11-28; First posted 2017-12-14 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: CD30-Positive Neoplastic Cells Present; Folliculotropic Mycosis Fungoides; Recurrent Mycosis Fungoides; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Mycosis Fungoides; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Sezary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Sezary Syndrome | interventions — Brentuximab Vedotin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brentuximab vedotin, lenalidomide) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 and lenalidomide PO QD on days 1-14. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Lenalidomide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: 914088-09-8; ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; Brentuximab Vedotin, cAC10-vcMMAE; SGN-35
Drug: Lenalidomide — Given PO
  Other Names: 191732-72-6; 3-(4-Amino-1-oxo-1,3-dihydro-2H-isoindol-2-yl)piperidine-2,6-dione; 703813; CC-5013; CC5013; CDC 501; Revlimid
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with brentuximab vedotin in treating patients with T-cell lymphomas that have come back or do not respond to treatment. Monoclonal antibodies, such as brentuximab vedotin, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving brentuximab vedotin and lenalidomide may work better in treating patients with T-cell lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD)/Recommended Phase 2 dose (RP2D) of brentuximab vedotin in combination with lenalidomide in patients with relapsed/ refractory cutaneous T-cell lymphoma (CTCL).

II. Assess safety and tolerability of brentuximab vedotin in combination with lenalidomide in patients with relapsed/ refractory CTCL.

SECONDARY OBJECTIVES:

I. Estimate the rate of objective global response that lasts at least 4 months (ORR4) , complete response (CR) rate, progression-free survival (PFS) of brentuximab vedotin in combination with lenalidomide in patients with relapsed/ refractory CTCL.

II. Estimate the rate and duration of clinically meaningful reduction in pruritus (CMRP).

III. Correlate response to baseline CD30 levels in tissue samples.

TERTIARY OBJECTIVES:

I. Estimate the response endpoints incorporating Lugano response criteria for patients with PET+ disease.

II. Explore temporal gene expression profile in skin/ blood samples that may predict response to combination therapy.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1 and lenalidomide orally (PO) once daily (QD) on days 1-14. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Registered into mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) program
* Women of childbearing potential: adhere to scheduled pregnancy testing as required in the Revlimid REMS program
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically confirmed cutaneous T-cell non-Hodgkin lymphoma (CTCL) per World Health Organization (WHO) classification 2016 including, mycosis fungoides (MF) or Sezary syndrome (SS); phase 1 : >= stage IIB OR >= stage IB-IIA folliculotropic/transformed MF; expansion cohort: >= stage IB

  * MF/SS stage of disease according to TNMB classification
  * SS is defined as meeting T4 plus B2 criteria; where the biopsy of erythrodermic skin may only reveal suggestive but not diagnostic histopathologic features, the diagnosis may be based on either node biopsy or fulfillment of B2 criteria
  * For MF where the histological diagnosis by light microscopic examination is not confirmed, diagnostic criteria that been recommended by the International Society for Cutaneous Lymphomas (ISCL) should be used
* Relapsed/refractory disease
* Failed >= 2 prior systemic therapies
* CD30-positivity by immunohistochemistry of >= 1%
* Measurable disease per modified Severity Weighted Assessment and/or Sezary count
* Fully recovered from acute toxicities (except alopecia) of all prior therapies to Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1
* May have received either brentuximab vedotin or lenalidomide/immunomodulatory imide drugs (IMiD) without dose modification/delay due to toxicity

  * IMiDs defined as thalidomide analogues
* If received prior brentuximab vedotin or lenalidomide, must be able to tolerate the dose level to which the participant will be enrolled to
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Absolute neutrophil count (ANC) >= 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Platelets >= 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Total bilirubin =< 1.5 X upper limit of normal (ULN) OR if Gilbert's syndrome =< 3.0 X ULN
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Aspartate aminotransferase (AST) =< 2 x ULN
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Alanine aminotransferase (ALT) =< 2 x ULN
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by WOCBP and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Stem cell transplantation
* Monoclonal antibody within 28 days prior to day 1 of protocol therapy
* Any systemic therapy, including monoclonal antibody within 28 days or 5 half-lives (whichever is shorter) of initiating day 1 of protocol therapy
* Any skin-directed therapy within 14 days prior to day 1 of protocol therapy
* Any radiation therapy within 21 days prior to day 1 of protocol therapy
* Immunosuppressive medication within 14 days prior to day 1 of protocol therapy; the following are exceptions to this criterion:

  * Intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection) and are on stable dose for at least 28 days
  * Systemic corticosteroids at physiologic doses of < 10 mg/day of prednisone or equivalent
* Live, attenuated vaccine within 30 days prior to day 1 of protocol therapy
* Disease free of prior malignancies for >= 5 years with the exception of:

  * Currently treated squamous cell and basal cell carcinoma of the skin, or
  * Carcinoma in situ of the cervix, or
  * Surgically removed melanoma in situ of the skin (stage 0) with histological confirmed free margins of excision , or
  * Prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) that has/have been surgically cured, or
  * Any other malignancy that has/have been curatively treated with surgery and/or localized radiation
* Allergic reaction/hypersensitivity to lenalidomide or history of anaphylactic shock to brentuximab vedotin in the past
* Female only: pregnant or breastfeeding
* Acute infection requiring systemic treatment
* Known history of human immunodeficiency virus (HIV) infection
* Active hepatitis B or C infection
* Central nervous system involvement by lymphoma, including leptomeningeal involvement
* History of progressive multifocal leukoencephalopathy (PML)
* Current peripheral neuropathy >= grade 2 or patients with the demyelinating form of Charcot-Marie-Tooth syndrome
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* History of vascular disease (e.g. deep vein thrombosis, stroke)
* Major surgery (as defined by the investigator) within the 28 days prior to day 1 of protocol therapy
* Incidence of gastrointestinal disease that may significantly alter the absorption of lenalidomide
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) assessed per CTCAE v4.0 | Up to 21 days

SECONDARY OUTCOMES:
Rate of objective global response defined as proportion of patients achieving complete response (CR)/partial response (PR) that lasts at least 4 months | At 4 months
  Will be estimated by the proportion of patients achieving a CR/PR that lasts at least 4 months, along with the 95% exact binomial confidence interval.
Complete response defined as proportion of patients achieving CR according to Olsen criteria | Up to 1 year
  Complete response rate will be estimated by the proportion of evaluable patients achieving CR, along with the 95% exact binomial confidence interval.
Progression free survival (PFS) according to Olsen criteria | From start of protocol treatment to first observation of disease relapse/ progression or death from any cause, whichever occurs first, assessed up to 1 year
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error.
Change in pruritus visual analogue scale (VAS) | Up to 1 year
  Pruritus visual analogue scale (VAS) is a horizontal 100mm long line on which the patients make a vertical mark to indicate their subjective assessment of pruritus intensity; the patients are informed that the scale represents no pruritus (0 points) to severe pruritus (100 points). Changes from baseline over time in pruritus VAS score will be assessed using descriptive statistics.
CD30 expression assessed by lymph node and/or skin biopsies via immunochemistry | Baseline
  Baseline CD30 levels in tissue samples by immunochemistry will be compared between responders and non-responders by Fisher's exact test. Log rank test will be used to explore the association between baseline CD30 levels in tissue samples with PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Zain, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States